CLINICAL TRIAL: NCT07083830
Title: A Phase I, Single Center Trial of Donor Extracorporeal Photopheresis (ECP) Treated Cell Infusion (ECP-DL) Plus Post-transplant ECP for the Prevention of Rejection in Living Donor Kidney Transplant Recipients
Brief Title: ECP-DL Cell Infusion for Induction in Living Donor Kidney (LDK) Transplants
Acronym: ECP
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Joseph Leventhal, Professor, Northwestern University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STU00222957
Record Dates: First submitted 2025-07-09; First posted 2025-07-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Kidney Transplant Failure and Rejection; Kidney Transplant; Complications
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ECP-DL Cell Therapy Arm (Experimental): Participants will receive escalating doses of ECP-DL (extracorporeal photopheresis-derived dendritic-like) cells starting on Day -7 prior to living donor kidney transplantation. The intervention aims to evaluate the safety and immunomodulatory effects of ECP-DL cell infusion in the context of renal transplantation.
  Interventions: Device: ECP-DL treated mononuclear cell infusion

INTERVENTIONS:
Device: ECP-DL treated mononuclear cell infusion — Participants in this study will undergo the infusion of donor white blood cells treated with ECP one week before their living donor kidney transplant, combined with standard of care antirejection medications. You will also then have ECP treatments using your own blood on two consecutive days once per month for 6 months. This combination is intended to cause your immune system to create a state called tolerance to the donor kidney. The ECP procedure has not been approved to prevent rejection after kidney transplant and the use of ECP to prevent rejection of transplanted organs is experimental, and is not a part of standard treatment which is based on the long term use of anti-rejection drugs such as tacrolimus (Prograf), everolimus, and prednisone.

SUMMARY:
This is a phase 1 trial, 36 month duration for subjects with end-stage renal disease (ESRD). The objectives of the trail are1) Determine the safety of ECP-DL cell infusion in living donor renal transplant recipients. 2) Determine rates of graft rejection and compare to historical controls.

One week prior to planned LDK transplant the donor and recipient pair will be seen for ECP-DL preparation and infusion. Donors will undergo one single unstimulated peripheral blood mononuclear cell collection using the THERAKOS® CELLEX® Photopheresis System; the cell product will then undergo ECP treatment to make ECP-DL, which will then be infused into the recipient. One week later, recipients (n=12) will undergo LDK transplant using standard of care maintenance immunosuppression without antibody induction therapy. Subsequent patients will receive cell infusions in escalating cell doses. A minimum of two months will be used as an interval between ECP-DL treatment in each tier. A staggered approach for moving to the next tier will be employed waiting no less than two months to ensure absence of adverse events using the following tier dosing schema:

Tier 1: 0.5 x 10^9 ECP-DL treated cells (n=4) Tier 2: 1 x 10^9 ECP-DL treated cells (n=4) Tier 3: 2 x 10^9 ECP-DL treated cells (n=4)

Following transplant, LDK recipients will undergo ECP using the Therakos system on two consecutive days per month for 6 months (12 treatments). Peripheral IV access will be used whenever possible.

ELIGIBILITY:
Inclusion Criteria:

* Recipient age ≥30 and less than 70 years old.
* Donor age ≥18 and ≤ 70 years old.
* Recipient of a first kidney transplant from a living unrelated or living related donor that is not HLA-identical to the donor.
* Donor willing to undergo cell collection for ECP-DL cell preparation and infusion.
* Donors will be screened and tested for HIV-1 (antigen and nucleic acid), HIV-2, hepatitis B virus (HBV, nucleic acid and surface and core antigen), hepatitis C virus (HCV, antigen and nucleic acid), Treponema pallidum (syphilis), West Nile Virus (WNV), and CJD (screening only). and tested for human T-lymphotropic virus types 1 and 2 (HTLV-1, HTLV-2) and CMV, in accordance with established UNOS guidelines for solid organ donors.
* Donors and recipients who test negative for TB using QuantiFERON gold assay.
* Must be willing and able to comply with protocol-required visit schedule and visit requirement.
* Patients who are single-organ recipients (kidney only).
* Women who are of childbearing potential must have a negative serum pregnancy test before transplantation and agree to use a medically acceptable method of contraception throughout the treatment period. Both male and female transplant recipients must agree to the use of highly effective birth control for 12 months following ECP-DL procedure. Individuals unwilling to do so will be excluded from study participation.
* Subjects are able to understand the consent form and give written informed consent.

Exclusion Criteria:

RECIPIENT

* Known sensitivity or contraindication to everolimus, tacrolimus, or psoralen.
* Aphakia.
* Has undergone splenectomy
* Patients with light-sensitive diseases including (but not limited to) systemic lupus erythematosus, porphyria cutanea tarda, erythropoietic protoporphyria, variegate porhyria, xeroderma pigmentosum, and albinism
* Patient with significant or active infection.
* Patients with a positive flow cytometric crossmatch using donor lymphocytes and recipient serum.
* Patients with PRA >80%
* Patients with current or historic donor specific antibodies
* Body Mass Index (BMI) of < 18 or > 40
* Patients who are pregnant or nursing mothers
* Patients whose life expectancy is severely limited by diseases other than renal disease
* Ongoing active substance abuse, drug or alcohol
* Major ongoing psychiatric illness or recent history of noncompliance
* Significant cardiovascular disease
* Malignancy within 3 years, excluding nonmelanoma skin cancers
* Subjects with cerebrovascular vascular disease with recent (< 6 months) stroke
* Serologic evidence of infection with HIV or HBVs Ag positive
* Recipient is EBV serologic negative
* Donor CMV serologic positive to recipient CMV serologic negative
* Recipient tests positive for HCV viral load by PCR
* Patients with a screening/baseline total white blood cell count < 4,000/mm3; platelet count < 100,000/mm3; triglyceride > 400 mg/dl; total cholesterol > 300 mg/dl
* Investigational drug within 30 days prior to transplant surgery
* Anti-T cell therapy within 30 days prior to transplant surgery
* Documented severe liver disease, defined as bridging fibrosis or cirrhosis on liver biopsy
* Poorly controlled diabetes, defined as HbA1c of > 8.0
* PT/INR > 2.0
* SBP < 90 or > 180mm Hg, HR > 120 or <50bpm, Temp > 99.5F on day of proposed ECP-DL procedure
* Patients receiving concomitant enteral or topical medical therapy with potentially photosensitizing effects

DONOR

* Lack of possible peripheral IV access (two access sites)
* Has undergone splenectomy
* Donor tests positive for HCV viral load by PCR
* PT/INR > 2.0; or known hyper or hypo coagulable disorders
* Hgb < 10.0
* platelet count < 100,000
* SBP < 90 or > 160mm Hg, HR > 120 or <50bpm, Temp > 99.5F on day of proposed ECP-DL procedure
* Donors who cannot tolerate extracorporeal volume during PBMC collection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2027-12-25 (Estimated); Study Completion 2028-08-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events Following Escalating Doses of ECP-DL Cells | From Day -7 (first ECP-DL infusion) through 24 months post transplant
  To determine the safety profile of escalating doses of ECP-DL cells administered to patients undergoing living donor kidney transplantation.

SECONDARY OUTCOMES:
Incidence of Transplant-Related Adverse Events | Baseline through 24 months post-transplant.
  To assess the frequency and type of adverse events associated with renal transplantation and immunosuppressive therapy.
Incidence and Severity of Infections | Baseline through 24 months post-transplant
  To evaluate the incidence, timing, and severity of bacterial, viral, and fungal infections post-transplant.
Changes in Peripheral Blood Lymphocyte Subpopulations | Baseline, Day 0, Day 7, Day 30, and Month 6
  To assess changes in lymphocyte subpopulations, including regulatory T cells and effector T cells, following ECP-DL infusion.
Change in Donor-Specific T Cell Response as Measured by Mixed Lymphocyte Reaction (MLR) and ELISPOT Assays | Baseline, Day 30, and Month 6
  Donor-specific hyporesponsiveness will be assessed by measuring the proliferation of recipient peripheral blood mononuclear cells (PBMCs) in response to donor antigens using Mixed Lymphocyte Reaction (MLR), and by quantifying interferon-gamma (IFN-γ) producing cells using ELISPOT assays. Results will be reported as stimulation index (SI) for MLR and spot-forming units (SFU) per 10^6 PBMCs for ELISPOT.
Quantitative Changes in Plasma and Urine Proteins Identified by Mass Spectrometry-Based Proteomic Analysis | Baseline, Day 30, and Month 6
  Blood and urine samples will be analyzed using mass spectrometry to measure changes in protein levels related to ECP-DL treatment and transplant outcomes. Protein levels will be reported using standard lab methods, and changes over time will be compared to identify significant differences.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Leventhal, MD, PhD, Principal Investigator — Northwestern University; Jennifer Schneiderman, MD, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago

IPD SHARING:
Plan to Share IPD: Undecided